CLINICAL TRIAL: NCT03009799
Title: Evaluation of the Efficacy and Safety of Iota-Carrageenan Eye Drops (NCX-4240) Versus Placebo in Patients With Adenoviral Conjunctivis
Brief Title: Efficacy and Safety of Iota-Carrageenan Eye Drops (NCX-4240)
Acronym: Goldeneye
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped following management decision
Sponsor: NicOx (Industry)
Collaborators: Iris Pharma (Industry); Theradis pharma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCX-4240-15001
Record Dates: First submitted 2016-12-12; First posted 2017-01-04 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Adenoviral Conjunctivitis
Keywords: adenoviral conjunctivis; iota-carrageenan
MeSH Terms: interventions — Carrageenan; Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eye drops containing Iota-Carrageenan (Active Comparator): Eye drops 3.2mg/ml
  Interventions: Drug: Iota-Carrageenan
- Ocular Lubricant Eye Drops (Placebo Comparator): Carmellose 0.5% sterile solution
  Interventions: Drug: Carmellose

INTERVENTIONS:
Drug: Iota-Carrageenan — One drop in each eye 8 times per day for 7 days (mandatory), then 4 to 8 times/day for the next 14 days until Day 21
  Other Names: NCX-4240
  Arms: Eye drops containing Iota-Carrageenan
Drug: Carmellose — 1 drop in each eye 8 times/day for 7 days (mandatory), then 4 to 8 times/day for the next 14 days until day 21
  Other Names: Placebo
  Arms: Ocular Lubricant Eye Drops

SUMMARY:
This clinical investigation aims at demonstrating that NCX-4240 is effective and safe in decreasing the number of days where adenoviral conjunctivis is detected in the eye and in reducing the duration and/or the severity of the signs and symptoms of adenoviral conjunctivis

DETAILED DESCRIPTION:
A multicenter, double masked, parallel, randomized 1:1 ratio clinical investigation comparing carrageenan eye drops (NCX 4240) versus placebo up to 21 days.

Total expected number of patients: 148

Randomization: patients will be randomized 1:1 between:

* Group A: eye drops containing iota-carrageenan (NCX 4240), 1 drop in each eye 8 times/day for 7 days (mandatory) then at least 4 to 8 times/day for the next 14 days until Day 21 or
* Group B: ocular lubricant eye drop (carmellose 0.5% sterile solution) 1 drop in each eye 8 times/day for 7 days (Mandatory), then 4 to 8 times/day for the next 14 days until Day 21.

ELIGIBILITY:
Inclusion Criteria:

* With uni-or bilateral acute adenoviral conjunctivis as diagnostised with adenoplus test
* Conjunctivis signs and symptoms in at least one eye AND positive adenoplus test in at least one eye whatever signs/symptoms and positive adenoplus test are from the same eye or not

Exclusion Criteria:

* Negative results with adenoplus test in both eyes
* a suspected bacterial, fungal, herpes, chlamydia or acanthamoeba co-infection, based on clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Viral eradication time NCX 4240 versus Placebo | 21 days
  Comparison in time to viral eradication in NCX-4240 and the placebo groups (when virus load is 0 or BLD - below the limit of detection) from the tears as measured by Polymerase Chain Reaction (PCR) at each visit.

SECONDARY OUTCOMES:
Quantitative PCR | 21 days
  1) Quantitative PCR (qPCR) results at all clinical investigation timepoints 4) Global patient discomfort with Likert 4 points scales: no discomfort - minimal - moderate - severe discomfort, assessed every day in the Patient's diary 5) Ocular signs as assessed by the investigators at each visit and for both eyes
Impact on daily activities | 21 days
  Impact of the disease on daily activities as measured by the patient daily with a 4 points Likert scale (no - minimal - moderate - severe) 5) Ocular signs as assessed by the investigators at each visit and for both eyes:
  * Degree of bulbar conjunctival injection/hyperaemia will be graded using the Mc Monnies grading scale for conjunctival hyperaemia
  * Other signs will be assessed with Likert 5 points scales: none - traces - mild - moderate - severe for chemosis (conjunctival edema), follicles, petechiae, and keratitis. Presence/absence of loco-regional lymphadenopathies will also be recorded
Patient discomfort | 21 days
  Global patient discomfort with Likert 4 points scales: no discomfort - minimal - moderate - severe discomfort, assessed every day in the Patient's diary
bulbar conjuntival infection | 21 days
  Ocular signs as assessed by the investigators at each visit and for both eyes: degree of bulbar conjunctival infection/hyperaemia will be graded using the McMonnies grading scale for conjunctival hypereaemia.
Other signs to be assessed | 21 days
  Ocular signs as assessed by the investigators at each visit and for both eyes:
  - Other signs will be assessed with Likert 5 points scales: none - traces - mild - moderate - severe for chemosis (conjunctival edema), follicles, petechiae, and keratitis.
loco-regional lymphadenopathies | 21 days
  Ocular signs as assessed by the investigators at each visit and for both eyes:
  Presence/absence of loco-regional lymphadenopathies
Ocular symptoms assessed by patients | 21 days
  Ocular symptoms as assessed by the patients in the patient diary: self-rated daily for 21 days: symptoms sum-score of pain, foreign body sensation, itchy eye(s), photophobia/light sensitivity, ocular secretions and eyelash matting. Assessments will be performed with Likert 5 points scales (none - traces - mild - moderate - severe).
Disease impact on daily activities | 21 days
  Impact of the disease on daily activities as measured by the patient daily with a 4 points Likert scale (no - minimal - moderate - severe)
Global patient discomfort | 21 days
  Global patient discomfort with Likert 4 points scales: no discomfort - minimal - moderate - severe discomfort, assessed every day in the Patient's diary
Adenoplus test results | 21 days
  AdenoPlus® test results, testing the studied eye at each post baseline visits.
Investigator's assessment of Membranes and pseudomembranes development | 21 days
  For both eyes: Development of membranes, pseudomembranes assessed by the investigator, incidence and severity (none - mild - moderate - severe)
Investigator's assessment of Membranes and pseudomembranes development | 21 days
  For both eyes: timing of occurrence if any
Investigator's assessment of Subepithelial Corneal Infiltrates development | 21 days
  For both eyes: Development of subepithelial corneal infiltrates (none - mild - moderate - severe) as assessed by the investigator
Investigator's assessment of Subepithelial Corneal Infiltrates development | 21 days
  For both eyes: Development of subepithelial corneal infiltrates: timing of occurrence as assessed by the investigator examination
Assessment of Incidence and severity of fellow eye signs and symptoms | 21 days
  If only one eye is affected (signs and symptoms) at baseline, assessment of the incidence and severity of the other eye signs and symptoms by the investigator
BCVA | 21 days
  Best corrected far Visual Acuity for both eyes (Day 1, 7, 14 and Day 21).
Global assessment of patient's satisfaction | 21 days
  Global assessment of the patient's satisfaction with the eye drops use with a 4 points Likert scale: poor, fair, good, excellent, will be performed at Day 7, 14 and 21
Adverse events | 21 days
  Safety parameters (Adverse Events/Serious Adverse Events)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Duquesroix, Study Director — NicOx
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided